CLINICAL TRIAL: NCT06171295
Title: Pharmacokinetics and Pharmacodynamics of Levobupivacaine During Continuous Caudal Epidural Analgesia in Newborns
Acronym: Levon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Eva Al Jamal, Head of clinical trial department, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Levon 1111111
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Analgesia
Keywords: C-CELA; newborn; analgesia; epidural; pain
MeSH Terms: conditions — Agnosia; Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: PK study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PK of Levobupivacain (Other): Newborns who received epidural anesthesia with Levobupivacain
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — The blood draws in specified time points

SUMMARY:
The goal of this clinical trial is to learn about the pharmacokinetics of levobupivacaine in newborns during the continus caudal epidural analgesia. This type of analgesia is used for severly ill newborns. There is a need to lower the opioid doses for this population who is undergoing the surgery due to the life threading indication. In some cases it is considered to use the epidural analgesia for the sake of the patient.

The main question is:

Is the commonly used dosing of 0,25% levobupivacaine in dose 0,2-0,3mg/kg/h the ideal dosing for these patients?

Is this type of dosing of epidural analgesia safe and effective for newborns?

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent of parent(s)/legal representative(s)
* Age younger than 45thweek of PMA
* Age older than 25thweek of PMA
* body weight (BW) more than 500g
* Previous or planned operation with great demand on POPM
* Other diseases demanding great POPM (even without any need of surgery)
* Vital functions of the patient will be stable and there will be no suspicion, that patient current condition might be worsen by insertion of c-CELA (every patient will be discussed with attending physician )

Exclusion Criteria:

* Decline of informed consent by parent(s) legal representative
* Age older than 45thweek of PMA
* Age younger than 25th week of PMA
* body weight (BW) lower than 500g
* Congenital malformation of caudal part of spine ( spina bifida occulta , meningocele, meningomyelocele)
* Disease or congenital malformation significantly restricting liver functions (Elevation of liver enzymes more than twice above the physiological range of the corresponding PMA)
* Disease or congenital malformation significantly restricting kidney functions (Elevation of urea and creatinine enzymes more than twice above the physiological range of the corresponding PMA)
* Clinical condition, which doesn't long-term POPM
* Meningism
* Patients with proven withdrawal syndrome caused by opiate administration
* High risk of bleeding during insertion (coagulopathy) or known administrated anticoagulants which might be still active in the time of insertion of c-CELA
* Substantial anemia (under 90g/l), which could lead to blood transfusion due to blood drawing
* frequent blood tests associated with the treatment of the patient(with blood samples necessary for the purposes of the study together), which would exceed maximum
* any hemodynamically unstable condition (for example septic shock)

Ages: 1 Hour to 5 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Safety | 144 hours
  AE, SAE monitoring, opioid intake monitoring
Effectivity | 144 hours
  Pain managment monitoring - Comfort Neo Scale

SECONDARY OUTCOMES:
Neurotoxicity | up to 5 years
  Follow up visits with basic neurology examination

CONTACTS AND LOCATIONS:
Overall Officials: Jan Šípek, Study Chair — University Hospital, Motol
Locations (1):
- University hospital Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No